CLINICAL TRIAL: NCT05629143
Title: Determining the Optimal Strategy for Stopping Chronic Proton Pump Inhibitor Therapy in Primary Care Patients: Impact of On-demand Use, Adjunctive Therapies and Antacids
Brief Title: Primary carE PPi dEprescRibing Trial
Acronym: PEPPER
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S64556
Record Dates: First submitted 2022-11-03; First posted 2022-11-29 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Heartburn; Dyspepsia; Reflux
Keywords: proton pump inhibitor
MeSH Terms: conditions — Heartburn; Dyspepsia; Gastroesophageal Reflux | interventions — Alginates

STUDY DESIGN:
Intervention Model Description: Evaluation of de-prescription strategies for PPIs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intermittent deprescribing strategy (Other): Classical approach for deprescribing of PPI based on Belgian Guidelines. In this study arm, the patients will keep the intake of their PPI but will decrease the use of PPI using a scheme where the PPI dose in reduced intermittently for one month. After one month in the intermittent deprescribing scheme, the patients will stop the use of PPI.
  Interventions: Procedure: de-prescription of PPI via intermittent scheme
- On-demand deprescribing strategy (Other): In this study arm, the patients will keep the intake of their PPI but will decrease the use of PPI in an on-demand bases for one month. The patient will only take the PPI when strictly needed because of symptoms. After one month in the on-demand PPI use, the patients will stop the use of PPI.
  Interventions: Procedure: de-prescription of PPI via on-demand scheme
- Replacement of PPI with alginate therapy (Other): In this study arm, the patient will stop the intake of the PPI band replace it with the use of an alginate for one month. After one month, the patient will stop the use of alginates.
  Interventions: Drug: Alginate

INTERVENTIONS:
Procedure: de-prescription of PPI via intermittent scheme — The patients will decrease their intake of PPIs via a de-prescription intermittent scheme. After one month, patients will stop their intake of PPI.
  Arms: Intermittent deprescribing strategy
Procedure: de-prescription of PPI via on-demand scheme — The patients will decrease their intake of PPIs via a de-prescription on-demand scheme. After one month, patients will stop their intake of PPI.
  Arms: On-demand deprescribing strategy
Drug: Alginate — The patients will stop their intake of PPIs and use alginate. After one month, patients will stop their intake of alginates.
  Arms: Replacement of PPI with alginate therapy

SUMMARY:
Proton pump inibitors (PPIs) is a class of medications that reduce the acid secretion in the stomach. These medications are very effective to relieve symptoms of acid reflux for a well-identified group of diseases and conditions.

Over the years, a major rise in use of these drugs has occurred. Convincing analyses reveal that a large share of this use occurs outside regular indications, at inappropriately elevated doses and prolonged treatment durations. Moreover, there are increasing concerns regarding potential adverse effects and the high cost associated with improper PPI use.

Guidelines propose to reduce chronic use of PPIs, but to date this has not generated a reduction in their application in clinical practice. One reason is the occurrence of a period of 2 weeks of increased acid secretion, with recurrence of symptoms, when these drugs are stopped after already a few weeks of usage (rebound effect). The best strategy to overcome this period of increased acid secretion and symptoms has not been established.

The PEPPER study will evaluate two different strategies to overcome the period of increased secretion when trying to interrupt chronic proton pump inhibitor therapy. The investigators will compare the success of stopping PPIs when these strategies are implemented, compared to a classical strategy of stopping after intermittent PPI intake. The strategies under evaluation are a period of non-daily intake of proton pump inhibitors (on-demand) before stopping, or the use of alternative methods to control gastric acidity and reflux (so-called alginates).

The investigators will evaluate the success rate of stopping chronic PPIs treatment with these approaches, compared to an interruption with intake of antacids. Patients will be followed up for 1 year after interruption of PPIs, and the level of symptom control, quality of life and healthcare costs will be evaluated at intervals.

The study will be conducted in patients from primary care practices with chronic PPIs intake outside of the established disease indications.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients are those of either gender, above the age of 18, eligible to give informed consent

* Based on indication: Patients on long-term (>12 weeks) chronic (daily) PPI use without therapy indication are eligible to participate.
* Based on dose:

  * Patients on a "maintenance" PPI dose are eligible for randomization. Maintenance dose is 20 mg of omeprazole, esomeprazole or pantoprazole daily or 15 mg of lansoprazole daily or 10 mg of rabeprazole daily.
  * Patients on a "healing" PPI dose (i.e. ≥40 mg esomeprazole, esomeprazole or pantoprazole or ≥30 mg of lansoprazole or ≥20 mg or rabeprazole daily) are also eligible, but need first to down-titrate their dose to "maintenance" dose before they can be considered for randomization.

Exclusion Criteria:

* Patients on short-term (<12 weeks) PPI therapy.
* Patients not on chronic PPI use (less than daily intake)
* Patients with established long-term indication such as the presence of a grade C, D oesophagitis, a peptic ulcer, Barrett's oesophagus or Zollinger-Ellison syndrome.
* Patients with chronic use of Gaviscon® or similar drugs based on magaldrate such as Riopan® and Gastricalm® (i.e. more than once a week for the last 2 months).
* Patients with chronic use of NSAIDs (i.e. two or more weekly doses).
* Patients with a history of gastric or oesophageal surgery.
* Patients with a major oesophageal disease such as achalasia, oesophageal spasm, or oesophageal involvement in systemic disease such as scleroderma or dermatomyositis.
* Patients with drug abuse and/or alcohol abuse
* Women who are pregnant or lactating
* Patients not able to understand or be compliant with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Succes of de-prescription strategy | 15 months
  percentage of randomized patients achieving successful therapeutic outcome at the end of the follow up period in each treatment group

SECONDARY OUTCOMES:
Use of PPI | 15 months
  Patient reported outcome The use of PPI will be reported by the patient at each study visit as adherence to the suggested treatment. As this information is considered as standard of care, this is the value that will be used for the analysis of this first key point that will be used for the assessment of the primary endpoint of the study.
  During follow up, patients taking at least one dose of PPIs weekly will be consider as active PPI users, and therefore a failure to this key indicator (result "0"). If patients report to have used a dose PPI less than 3 times in a month, this subject will not be consider as clinical relevant users, and therefore the key indicator result is positive and "1".
Treatment satisfaction | 15 months
  Patient reported outcome Scale title:treatment satisfaction scale Question to assess treatment satisfaction is: "How satisfied or dissatisfied are you with the control of your symptoms with the current treatment?" Minimum and maximum values: seven-point bipolar scale from 'Extremely Satisfied' (score 7) to 'Extremely Dissatisfied' (score 1) Higher scores mean: better outcome
Willingness to continue with the current treatment | 15 months
  Patient reported outcome To assess willingness to continue to current treatment regimen, the following question will be used: "Would you be willing to continue the current treatment for the next month?"

OTHER OUTCOMES:
Economic impact of PPI deprescribing | 15 months
  Title: Health resource utilisation questionnaire Minimum and maximum values: yes or no questions (1 or 0) regarding use health resource use Higher scores mean: worst outcome as this is related to more expences due to health issues
Predictor of success - Predictive value of the symptom pattern | 15 months
  Patient reported outcome questionnaire title:esophageal and gastric symptoms questionnaire Min and max values: varies based on the question to presence of a symptom: yes-no questions and the severity of symptoms with higher scores for more severe symptoms.
  Higher scores means worst outcome as symptoms are more present and more severe.
Predictive value of demographic variables | 15 month
  Demographic assessment with patients questionnaires
Predictive value of number of co-morbidities to stop PPIs use | 15 months
  Co-morbidities assessment via GP via eCRF The investigator will evaluate if increased number of co-morbidities is a predictor for lower likelihood to succeed a the treatment to decrease the use of PPI.
Predictive value of number of previous failed attempts to stop PPIs use | 15 months
  Assessment via eCRF via GP medical assessment The investigator will evaluate if the number of previous failed attempts to stop PPIs use is a predictor for lower likelihood to succeed a the treatment to decrease the use of PPI.
Predictive value of gastrin level | 15 months
  Blood sample at baseline and after 1 year follow-up
Predictive value of the level of patients' motivation to stop PPIs use | 15 months
  Patient reported outcome on motivation during the study title: Motivational visual analogue scale Max-min scores: 100-0 from "extremely motivated" to "no motivation" Higher scores: good outcome The investigator will evaluate if the level of motivation to stop PPIs use is a predictor for likelihood to succeed a the treatment to decrease the use of PPI.
Work productivity impact of PPI deprescribing | 15 months
  title: Work productivity impact questionnaire (WPAI) Max-Min scores: yes/no questions (1/0) and number of hours worked per week (scores: 0 to 150) Higer scores= good outcome, as the patients feels good to work and be productive
Number of participants using rescue therapy | 15 months
  Assessment via questionnaire in ePRO

CONTACTS AND LOCATIONS:
Locations (1):
- Jan Tack, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
no individual data sharing